CLINICAL TRIAL: NCT00409916
Title: Prevention of Heart Failure Events With Impedance Cardiography Testing (PREVENT-HF)
Brief Title: PREVENT-HF: Prevention of Heart Failure Events With Impedance Cardiography Testing
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CardioDynamics (Industry)
Responsible Party: Rhonda Rhyne, President, CardioDynamics
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 06001-M2-124-1-3
Record Dates: First submitted 2006-12-08; First posted 2006-12-12 (Estimated); Last update posted 2009-06-03 (Estimated); Status verified 2009-06

CONDITIONS: Heart Failure, Congestive
Keywords: chronic heart failure; heart failure; congestive heart failure; impedance cardiography; ICG; transthoracic electrical bioimpedance; non-invasive; TEB
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Care Arm (Placebo Comparator): In the Standard Care Arm, the treating clinician will adjust therapy according only to the clinical assessment of signs and symptoms of heart failure since the ICG information is blinded to the treating clinician.
  Interventions: Device: BioZ Dx
- ICG Arm (Active Comparator): In the ICG Arm, the treating clinician will adjust therapy according to the clinical assessment of signs and symptoms of heart failure, in addition to the ICG hemodynamic information obtained from the printed report.
  Interventions: Device: BioZ Dx

INTERVENTIONS:
Device: BioZ Dx

SUMMARY:
The purpose of this study is to determine whether outpatient therapeutic management guided by impedance cardiography (ICG), in addition to standard clinical assessment, will result in a longer time in days to the first heart failure hospitalization than therapy guided by clinical assessment alone.

DETAILED DESCRIPTION:
The course of patients with chronic heart failure is marked by periodic episodes of clinical decompensation that not only impair the quality of life and may be fatal but also consume substantial health care resources, primarily due to the costs of hospitalization. Heart failure management programs have been developed to reduce the frequency and severity of these clinical events, but their effectiveness may be limited by physicians' difficulty in identifying patients at imminent risk. Reliable prediction of these events may afford physicians the opportunity to intervene aggressively and potentially minimize the need for hospitalization or the risk of a serious adverse outcome.

Noninvasive impedance cardiography (ICG) is a simple test that utilizes changes in thoracic electrical impedance to measure thoracic fluid content, changes in the duration of cardiac ejection and the velocity of blood flow within the aorta. ICG has been used to estimate cardiac output and cardiac filling pressure in patients with or without heart failure (HF).

PREVENT-HF is a randomized prospective study being conducted at up to 35 experienced investigative centers from the United States, Canada, and Europe. Subjects will be enrolled within 4-12 days of a discharge from a hospitalization for exacerbation of heart failure, with screening procedures to occur prior to the enrollment. Following enrollment, subjects will be randomized in a 1:1 ratio to outpatient management by either clinical assessment (Standard Care Arm) or ICG in addition to clinical assessment (ICG Arm) during the enrollment visit. ICG variables will be collected in all subjects but will be blinded in the Standard Care Arm. Each subject's study participation will last for a minimum of 24 weeks and a maximum of 52 weeks post-discharge. Four weeks after hospital discharge, subjects will visit the clinic. Remaining study visits will occur every four weeks thereafter until the subject has completed the 52-week visit or until the subject has experienced a hospitalization that has been adjudicated by the Clinical Events Committee as being a heart failure hospitalization.

In the PREDICT study, a composite ICG score was the most powerful predictor of a short-term HF event when compared to standard clinical variables. This composite ICG score is provided for subjects in the PREVENT-HF ICG Arm. If the score indicates a subject is at a higher risk for a short-term HF event, clinicians will be required to intervene. Clinicians may intervene if indicated by the subject's clinical status for an intermediate-risk score, and intervention is not recommended based on the ICG score for lower-risk scores. Compliance to these guidelines will be tracked.

ELIGIBILITY:
Inclusion Criteria:

* Discharge within 12 days from a hospitalization with the primary diagnosis of heart failure
* Age 18 years or older
* Chronic heart failure of at least 2 months' duration due to an ischemic or nonischemic etiology
* Receiving medications for heart failure that are considered (in the judgment of their physician) as being appropriate for their clinical status
* Able to acquire data successfully with the BioZ device
* Able and willing to provide written informed consent

Exclusion Criteria:

* Height < 48 inches or > 90 inches (< 120 cm or > 230 cm); weight < 67 lbs or > 341 lbs (<30 kg or >155 kg)
* Acute heart failure due to myocarditis, cor pulmonale, congenital heart disease, constrictive pericarditis, or hypertrophic, restrictive or obstructive cardiomyopathy
* Presence of severe aortic regurgitation
* Acute coronary syndrome (myocardial infarction or unstable angina) or coronary revascularization procedure (coronary bypass surgery or angioplasty) within 2 months
* History of resuscitated sudden death, ventricular fibrillation, or hemodynamically destabilizing VT unless treated with a properly functioning ICD
* One or more episodes of ventricular fibrillation or hemodynamically destabilizing ventricular tachycardia within the previous 30 days
* Second degree - Mobitz Type II or third degree heart block, unless treated with a cardiac pacemaker
* Implantation of a left ventricular assist device, hemodynamic monitor, activated minute ventilation pacemaker, or biventricular pacemaker (cardiac resynchronization therapy) with the V-to-V interval set at more than 5 milliseconds offset
* Implantation of a CRT (cardiac resynchronization therapy) device within the previous 30 days
* Planned implantation of a CRT within the next 6 months
* Clinician use of intrathoracic impedance data from an implanted pacemaker with this capability
* Participation in a transtelephonic or internet-based formal monitoring program
* Most recent serum creatinine > 3 mg/dl; any liver function test (ALT, AST or bilirubin) > 3 times the upper limit of normal; chronic dialysis; or chronic ultrafiltration
* Plan to serially monitor B-type natriuretic peptide (BNP) or N-terminal prohormone of B-type natriuretic peptide (NT-proBNP) as part of outpatient management
* Post-discharge management with outpatient infusions
* Pulmonary disease sufficient to significantly limit exercise or requiring long-term treatment with oral corticosteroids
* Known hypersensitivity or allergies to sensor gel or adhesive; skin lesions that prohibit adequate sensor placement
* Women known to be pregnant or who are planning to become pregnant in the next 12 months
* Current participation in other investigational drug or device protocols, with the exceptions of registries and subjects in long-term safety follow-up with no active treatment for at least 60 days
* Subjects with a disorder other than heart failure that might be expected to compromise their survival within the next 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2007-01; Primary Completion 2011-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Time in days to first heart failure hospitalization following study enrollment compared between study arms

SECONDARY OUTCOMES:
Time in days to the first heart failure hospitalization or all-cause death between study arms (a composite endpoint without weighting)
Number of total heart failure hospitalizations compared between study arms
Improvement in Quality of Life scores compared between study arms at 4, 12, 24, and 52 weeks versus baseline
Improvement in Patient Global Assessment compared between study arms at 4, 12, 24, and 52 weeks versus baseline
NYHA functional class at 4, 12, 24, and 52 weeks versus baseline in the ICG study arm
Prognostic capability of the blinded BioZ score in the Standard Care arm for short-term heart failure events.

CONTACTS AND LOCATIONS:
Overall Officials: Milton Packer, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (3):
- United States (3):
  - Sutter Memorial Hospital, Sacramento, California
  - Scripps Clinic, San Diego, California
  - University of California at San Diego, San Diego, California

REFERENCES:
- [Background] Packer M, Abraham WT, Mehra MR, Yancy CW, Lawless CE, Mitchell JE, Smart FW, Bijou R, O'Connor CM, Massie BM, Pina IL, Greenberg BH, Young JB, Fishbein DP, Hauptman PJ, Bourge RC, Strobeck JE, Murali S, Schocken D, Teerlink JR, Levy WC, Trupp RJ, Silver MA; Prospective Evaluation and Identification of Cardiac Decompensation by ICG Test (PREDICT) Study Investigators and Coordinators. Utility of impedance cardiography for the identification of short-term risk of clinical decompensation in stable patients with chronic heart failure. J Am Coll Cardiol. 2006 Jun 6;47(11):2245-52. doi: 10.1016/j.jacc.2005.12.071. Epub 2006 May 15. PMID 16750691